CLINICAL TRIAL: NCT02185599
Title: IMproved PRactice Outcomes and Value Excellence in Colposcopy
Acronym: IMPROVE-COLPO
Status: Completed | Type: Observational
Sponsor: DySIS Medical Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: IMPROVE-100
Record Dates: First submitted 2014-07-04; First posted 2014-07-09 (Estimated); Last update posted 2020-03-13 (Actual); Status verified 2020-03

CONDITIONS: High Grade Cervical Intraepithelial Neoplasia
Keywords: colposcopy; CIN; cervical neoplasia; cervical dysplasia; cervical cancer; CIN2+
MeSH Terms: conditions — Uterine Cervical Dysplasia; Uterine Cervical Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Colposcopy with DySIS: The prospective arm will recruit patients referred for colposcopy and will be examined using DySIS.
  Interventions: Device: DySIS
- Standard colposcopy: The retrospective arm will collect historical data from colposcopy examinations performed using a standard colposcope.

INTERVENTIONS:
Device: DySIS — Colposcopy performed with the DySIS digital colposcope
  Groups: Colposcopy with DySIS

SUMMARY:
The study will observe and quantify shifts in colposcopy practice and outcome improvements in U.S. community-based cervical screening colposcopy examinations after the introduction of the DySIS colposcope with Advanced Cervical Scan.

The study will collect colposcopy data across multiple sites in two arms; a prospective arm, with DySIS being used for the examination and a retrospective arm, with data retrieved from patient charts.

DETAILED DESCRIPTION:
Each site will contribute data to both arms; the study will collect data on demographics, disease yield, number of biopsies and treatment decisions. Study subjects will receive standard of care procedures and management.

Prospective data will be collected at colposcopy examinations performed using the DySIS digital colposcope on consecutive patients that have been referred for colposcopy after a positive screening test. Retrospective data on colposcopy examinations performed using a standard colposcope will be collected from patient medical records, to capture standard practice to-date as a control for comparisons. The retrospective data will be collected from consecutive examinations performed by the providers participating in the prospective arm and for the preceding year.

ELIGIBILITY:
Inclusion Criteria:

1. Females 21 years or older
2. Able to give informed consent
3. Referred for colposcopy with a screening test result that indicates the need for a colposcopy, based on guidelines and practice:

   * HSIL, ASC-H, LSIL cytology
   * 2x ASC-US cytology (25 or above)
   * 2x/3x LSIL/ASC-US cytology (21-24)
   * ASC-US pap and hrHPV cotest/reflex
   * HPV 16/18 primary screening (≥25)
   * ASC-US pap after hrHPV
   * hrHPV x2 (≥30)
   * HPV16 or 16 after negative cytology/hrHPV (≥30)
   * Follow-up of CIN2/3 biopsy (younger women)
   * hrHPV and/or ≥ASC-US pap post-excision

Exclusion Criteria:

1. Previous hysterectomy, previous/current chemotherapy, radiation treatment for cervical neoplasia or other concurrent cancer
2. Pregnancy
3. Known human immunodeficiency virus (HIV) infection or acquired immune deficiency syndrome (AIDS)
4. Referred for vulva/vaginal disease

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women referred for colposcopy after an abnormal screening test for prevention of cervical cancer
Sampling Method: Probability Sample
Enrollment: 7555 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2017-10-09 (Actual); Study Completion 2017-10-09 (Actual)

PRIMARY OUTCOMES:
Number of subjects diagnosed with CIN2+ cervical lesions | At time of colposcopy
  Changes in number of subjects diagnosed with CIN2+ cervical lesions

CONTACTS AND LOCATIONS:
Locations (46):
- United States (46):
  - Arizona Oncology, Scottsdale, Arizona
  - Unified Women's Clinical Research-Gainesville, Gainesville, Florida
  - North Florida OB GYN Associates, PA, Jacksonville, Florida
  - Osceola Ob-Gyn, PA, Kissimmee, Florida
  - Unified Women's Clinical research-Alpharetta, Alpharetta, Georgia
  - Unified Women's Clinical Research-Atlanta, Atlanta, Georgia
  - Northeast Georgia Physicians Group- Heritage, Gainesville, Georgia
  - Lakeside Ob/Gyn-Northeast Georgia Physician Group, Hoschton, Georgia
  - Nye Partners in Women's Health, Chicago, Illinois
  - Advocate Illinois Masonic Medical Center - Creticos Cancer Center, Chicago, Illinois
  - Midwest Center for Women's Healthcare, Elgin, Illinois
  - Advanced Women's Healthcare Specialists, SC, Elk Grove Village, Illinois
  - Providea Health Partners, LLC, Evergreen Park, Illinois
  - Women's Wellness World, Hazel Crest, Illinois
  - Women's Healthcare of Illinois, Mokena, Illinois
  - The Advanced Gynecologic Surgery Institute, Naperville, Illinois
  - Women's Center for Health, Naperville, Illinois
  - Southwest Women's Healthcare Associates, Olympia Fields, Illinois
  - Hinsdale & Oak Brook Women's Clinic, Willowbrook, Illinois
  - OB-GYN Associates, Cedar Rapids, Iowa
  - Margaret A. Smollen, MD, PC, Iowa City, Iowa
  - Brodsky & Taylor, PLC, Ferndale, Michigan
  - Downriver Obstetrics & Gynecology, Trenton, Michigan
  - NJ Gynecological Institute, Hackensack, New Jersey
  - Women's Healthcare of Princeton, LLC, Princeton, New Jersey
  - New Beginnings, OB/GYN, Springfield, New Jersey
  - Dr Gregory Shifrin, OB/GYN, PC, Brooklyn, New York
  - Unified Women's Clinical Research-Cary, Cary, North Carolina
  - Unified Women's Clinical Research-Greensboro, Greensboro, North Carolina
  - Unified Women's Clinical Research- Central Carolina, Greensboro, North Carolina
  - Lyndhurst Clinical Research- Mt Airy, Mount Airy, North Carolina
  - Lyndhurst Clinical Research, Winston-Salem, North Carolina
  - The Women's Center at Southview, Dayton, Ohio
  - Physicians & Surgeons for Women, Inc, Springfield, Ohio
  - The University of Toledo, Toledo, Ohio
  - Austin Area OB-Gyn, Austin, Texas
  - Coastal Bend Women's center, Corpus Christi, Texas
  - Laura Bradford, MD, Fort Worth, Texas
  - Las Colinas OBGyn, Irving, Texas
  - MacArthur OB/GYN, Irving, Texas
  - Advanced Women's Wellness, Katy, Texas
  - Zeid Women's Health Center, Longview, Texas
  - Craig Ranch Ob/Gyn, McKinney, Texas
  - Advanced Ob-Gyn Associates, Richardson, Texas
  - Dr DeLeon's Women's Healthcare, Rowlett, Texas
  - Piedmont Preferred Women's Healthcare Associates, Ridgeway, Virginia